CLINICAL TRIAL: NCT00901576
Title: A Phase 1, Open-label, Randomized, Three-period Crossover Drug Interaction Study Evaluating the Pharmacokinetic Profiles of SPD503 and CONCERTA, Administered Alone and in Combination in Healthy Adult Volunteers
Brief Title: A Drug Interaction Study of SPD503 and Concerta Administered Alone and In Combination in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD503-114
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Guanfacine; Methylphenidate

ARMS (3):
- SPD503 (Experimental)
  Interventions: Drug: SPD503
- Concerta (Active Comparator)
  Interventions: Drug: Concerta
- SPD503 + Concerta (Active Comparator)
  Interventions: Drug: SPD503 + Concerta

INTERVENTIONS:
Drug: SPD503 — SPD503 (guanfacine hydrochloride) extended-release 4 mg orally administered tablets
  Other Names: Intuniv
  Arms: SPD503
Drug: Concerta — CONCERTA (methylphenidate HCl) extended-release 36 mg orally administered tablets.
  Arms: Concerta
Drug: SPD503 + Concerta — SPD503 4 mg + CONCERTA 36 mg orally administered tablets (taken together).
  Arms: SPD503 + Concerta

SUMMARY:
This is a drug-drug interaction study; the purpose of this study is to examine the pharmacokinetics (levels of drug in the blood) of SPD503 (guanfacine hydrochloride) and Concerta (methylphenidate HCl) when given alone, and in combination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be normal healthy adult volunteers with no significant abnormalities in medical history, physical exam, vital signs or lab evaluations at the screening visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-05-18 (Actual); Primary Completion 2009-07-06 (Actual); Study Completion 2009-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Advanced Biomedical Research, Inc., Hackensack, New Jersey, United States

REFERENCES:
- [Result] Roesch B, Corcoran M, Haffey M, Stevenson A, Wang P, Purkayastha J, Martin P, Ermer J. Pharmacokinetics of coadministration of guanfacine extended release and methylphenidate extended release. Drugs R D. 2013 Mar;13(1):53-61. doi: 10.1007/s40268-013-0009-5. PMID 23519656
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consists of 3 regimens: SPD503 (extended-release guanfacine HCl) single 4 mg dose, Concerta (extended-release methylphenidate HCl) single 36 mg dose, and SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered. Each dosing regimen is separated by a washout period and performed in 6 different dosing sequences.
Groups:
- SPD503 First, Then Concerta, Then SPD503 + Concerta: SPD503 single 4 mg dose in first intervention, washout, Concerta single 36 mg dose in second intervention, washout, SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered in third intervention
- SPD503 First, Then SPD503 + Concerta, Then Concerta: SPD503 single 4 mg dose in first intervention, washout, SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered in second intervention, washout, Concerta single 36 mg dose in third intervention
- Concerta First, Then SPD503, Then SPD503 + Concerta: Concerta single 36 mg dose in first intervention, washout, SPD503 single 4 mg dose in second intervention, washout, SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered in third intervention
- Concerta First, Then SPD503 + Concerta, Then SPD503: Concerta single 36 mg dose in first intervention, washout, SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered in second intervention, washout, SPD503 single 4 mg dose in third intervention
- SPD503 + Concerta First, Then SPD503, Then Concerta: SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered in first intervention, washout, SPD503 single 4 mg dose in second intervention, washout, Concerta single 36 mg dose in third intervention
- SPD503 + Concerta First, Then Concerta, Then SPD503: SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered in first intervention, washout, Concerta single 36 mg dose in second intervention, washout, SPD503 single 4 mg dose in third intervention
Period: First Intervention
Arm/Group | SPD503 First, Then Concerta, Then SPD503 + Concerta | SPD503 First, Then SPD503 + Concerta, Then Concerta | Concerta First, Then SPD503, Then SPD503 + Concerta | Concerta First, Then SPD503 + Concerta, Then SPD503 | SPD503 + Concerta First, Then SPD503, Then Concerta | SPD503 + Concerta First, Then Concerta, Then SPD503
Started | 6 | 7 | 7 | 6 | 6 | 6
Completed | 6 | 7 | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | SPD503 First, Then Concerta, Then SPD503 + Concerta | SPD503 First, Then SPD503 + Concerta, Then Concerta | Concerta First, Then SPD503, Then SPD503 + Concerta | Concerta First, Then SPD503 + Concerta, Then SPD503 | SPD503 + Concerta First, Then SPD503, Then Concerta | SPD503 + Concerta First, Then Concerta, Then SPD503
Started | 6 | 7 | 7 | 6 | 6 | 6
Completed | 6 | 7 | 7 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | SPD503 First, Then Concerta, Then SPD503 + Concerta | SPD503 First, Then SPD503 + Concerta, Then Concerta | Concerta First, Then SPD503, Then SPD503 + Concerta | Concerta First, Then SPD503 + Concerta, Then SPD503 | SPD503 + Concerta First, Then SPD503, Then Concerta | SPD503 + Concerta First, Then Concerta, Then SPD503
Started | 6 | 7 | 7 | 6 | 6 | 6
Completed | 5 | 7 | 7 | 5 | 6 | 5
Not Completed | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | SPD503 First, Then Concerta, Then SPD503 + Concerta | SPD503 First, Then SPD503 + Concerta, Then Concerta | Concerta First, Then SPD503, Then SPD503 + Concerta | Concerta First, Then SPD503 + Concerta, Then SPD503 | SPD503 + Concerta First, Then SPD503, Then Concerta | SPD503 + Concerta First, Then Concerta, Then SPD503
Started | 5 | 7 | 7 | 5 | 6 | 5
Completed | 5 | 7 | 7 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | SPD503 First, Then Concerta, Then SPD503 + Concerta | SPD503 First, Then SPD503 + Concerta, Then Concerta | Concerta First, Then SPD503, Then SPD503 + Concerta | Concerta First, Then SPD503 + Concerta, Then SPD503 | SPD503 + Concerta First, Then SPD503, Then Concerta | SPD503 + Concerta First, Then Concerta, Then SPD503
Started | 5 | 7 | 7 | 5 | 6 | 5
Completed | 5 | 7 | 7 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD503 First, Then Concerta, Then SPD503 + Concerta | SPD503 First, Then SPD503 + Concerta, Then Concerta | Concerta First, Then SPD503, Then SPD503 + Concerta | Concerta First, Then SPD503 + Concerta, Then SPD503 | SPD503 + Concerta First, Then SPD503, Then Concerta | SPD503 + Concerta First, Then Concerta, Then SPD503 | Total
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6 | 6 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 7 | 6 | 6 | 6 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.54) | 32.6 (6.70) | 32.1 (8.01) | 31.5 (8.41) | 29.8 (2.64) | 30.3 (5.68) | 30.8 (6.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 1 | 1 | 2 | 9
  Male | 5 | 6 | 4 | 5 | 5 | 4 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 7 | 6 | 6 | 6 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: Pharmacokinetic Population (PKP) consists of all subjects in the Safety Population who had evaluable concentration-time profiles for guanfacine or d-methylphenidate. The Safety Population consists of all subjects who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- SPD503 Alone: Single 4 mg dose of extended-release Guanfacine HCl
- SPD503 + Concerta: SPD503 (single 4 mg dose) + Concerta (single 36 mg dose) coadministered
Arm/Group | SPD503 Alone | SPD503 + Concerta
Number analyzed (Participants) | 37 | 36
ng/ml | 2.6 (0.9) | 2.7 (0.9)

2. Primary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | SPD503 Alone | SPD503 + Concerta
Number analyzed (Participants) | 33 | 34
ng*h/ml | 96.5 (37.3) | 106.7 (39.9)

3. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SPD503 Alone | SPD503 + Concerta
Number analyzed (Participants) | 37 | 36
hours | 8.1 (8.1) | 8.7 (6.3)

4. Primary Outcome: Time of Plasma Half-Life(T 1/2) of Guanfacine
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SPD503 Alone | SPD503 + Concerta
Number analyzed (Participants) | 33 | 34
hours | 20.4 (7.9) | 22.7 (10.6)

5. Primary Outcome: Cmax of d-Methylphenidate
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Concerta Alone: Single 36 mg dose of extended-release Methylphenidate HCl
Arm/Group | Concerta Alone | SPD503 + Concerta
Number analyzed (Participants) | 38 | 37
ng/ml | 9.9 (2.8) | 9.5 (2.9)

6. Primary Outcome: AUC of d-Methylphenidate
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Concerta Alone | SPD503 + Concerta
Number analyzed (Participants) | 32 | 32
ng*h/ml | 102.8 (34.6) | 100.5 (33.0)

7. Primary Outcome: Tmax of d-Methylphenidate
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Concerta Alone | SPD503 + Concerta
Number analyzed (Participants) | 38 | 37
hours | 6.9 (1.0) | 7.4 (1.3)

8. Primary Outcome: T 1/2 of d-Methylphenidate
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 30, 48 and 72 hours post-dose
Population: PKP
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Concerta Alone | SPD503 + Concerta
Number analyzed (Participants) | 32 | 32
hours | 3.9 (0.7) | 4.1 (0.6)

ADVERSE EVENTS:
Description: Safety Population (SP) consisted of all subjects who received at least 1 dose of study drug and had at least 1 post-dose safety assessment
Arm/Group | SPD503 Alone | Concerta Alone | SPD503 + Concerta
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 6/37 | 8/38 | 4/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 Alone (N=37) | Concerta Alone (N=38) | SPD503 + Concerta (N=37)
Orthostatic syncope (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 Alone (N=37) | Concerta Alone (N=38) | SPD503 + Concerta (N=37)
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1
Dizziness postural (Nervous system disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.